CLINICAL TRIAL: NCT02617641
Title: Evaluation of a Web-Based Tailored Nursing Intervention (TAVIEenM@RCHE) Aimed at Increasing Walking in Patients After an Acute Coronary Syndrome: A Multicenter Randomized Controlled Trial
Brief Title: A Web-Based Tailored Nursing Intervention to Increase Walking in Patients After an Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Cossette, Ph.D., Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-1887
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Secondary Prevention; Walking; Health Behavior; Internet; eHealth; Computer-Assisted Instruction; Multicenter Study; Randomized Controlled Trial; Intervention Studies; Motivation; Self Efficacy; Theory, Nursing; Theory, Psychological; Nursing Research
MeSH Terms: conditions — Acute Coronary Syndrome; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAVIEenM@RCHE intervention (Experimental): The experimental group will receive a web-based tailored nursing intervention. Between 3 and 4 sessions of 15 to 25 minutes each are completed within 4 weeks. A booster session is delivered at 8 weeks post randomization.
  Interventions: Behavioral: TAVIEenM@RCHE
- Publicly available websites (Active Comparator): The control group will receive hyperlinks to four publicly available websites and one online booklet on the topic of walking.
  Interventions: Behavioral: Publicly available websites

INTERVENTIONS:
Behavioral: TAVIEenM@RCHE — The intervention goal is to increase up to 150 minutes per week of moderate-intensity physical activity through walking. The intervention is underpinned by Strengths-Based Nursing Care that specifies nursing values, and by Self-Determination Theory that specifies variables to tailor the intervention. The four intervention strategies are: 1) Providing information and feedback, 2) Exploring reasons to build motivation, 3) Exploring strengths to build confidence (self-efficacy), and 4) Developing an action plan to maintain motivation and confidence (self-efficacy). The TAVIE system platform is designed to provide a fully automated, easy to navigate website, and the main mode of delivery is video clips of a 'virtual nurse' who presents the tailored intervention content.
  Arms: TAVIEenM@RCHE intervention
Behavioral: Publicly available websites — * Le Programme de marche (Institut de Cardiologie de Montréal)
  * L'activité physique (Institut de Cardiologie de Montréal)
  * L'activité physique (Fondation des maladies du cœur et de l'AVC)
  * Directives canadiennes en matiére d'activité physique à l'intention des adultes âgés de 65 ans et plus (Société Canadienne de Physiologie de l'exercice)
  * Directives canadiennes en matière d'activité physique à l'intention des personnes âgées de 65 et plus (ParticipACTION)
  Arms: Publicly available websites

SUMMARY:
Acute coronary syndromes (ACS) are one of the leading causes of coronary artery disease mortality, and among the top reasons for health care utilization in Canada. Physical activity counselling is a core component of secondary prevention interventions because increased physical activity is associated with reduced mortality risk, improved quality of life, reduced coronary risk factors, and reduced health care utilization. Despite these health benefits, between 40% and 60% of patients after an ACS event are insufficiently active. Web-based interventions offer innovative alternatives for intervention delivery via the Internet in secondary prevention. However, there is a paucity of randomized controlled trials testing, in ACS patients, computer-tailored interventions that include videos within the tailored algorithm. The purpose of this multicenter randomized controlled trial is to test a web-based intervention, TAVIEenM@RCHE, that uses tailored-videos of a nurse, the 'virtual nurse', aimed at increasing physical activity through walking in ACS patients.

DETAILED DESCRIPTION:
After baseline data is collected, the participants (N = 148) will be randomized to either one of two groups: 1) access to the 4-week TAVIEenM@RCHE intervention with an additional "booster" at 8 weeks (experimental group) or 2) access to a list of publicly available websites (control group). Participants will be included if they report insufficient levels of physical activity prior hospitalization, and they have no serious medical conditions impeding adherence to moderate-intensity physical activity. Data collection will occur at recruitment (in-hospital), at baseline (home 3 weeks post-hospital discharge), and at 5 and 12 weeks post baseline. The data analysis will be consistent with intention-to-treat principles. Baseline characteristics will be compared using descriptive statistics to identify trends in group imbalances. For the analysis of the primary outcome of change in steps per day between baseline and 12 weeks, and the secondary outcome of change in steps per day between baseline and 5 weeks, a repeated measures ANCOVA model will compare the adjusted differences between the experimental and control groups at a significance of 0.05. For the analysis of the two secondary outcomes of change in energy expenditure in walking and in moderate-intensity physical activity between baseline and 5 weeks, and between baseline and 12 weeks, a repeated measures MANCOVA model will compare the adjusted differences between the experimental and control groups at a significance of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Discharged 3 weeks home post ACS-related hospitalization.
2. No serious medical condition exists that would impede adhering to moderate-intensity physical activity. Medical conditions include, for instance, incapacitating chronic pain, paralysis, equilibrium problems, diabetic ulcers, fluid restrictions, dyspnea, home oxygen dependency, cancer and others. Also, no environmental restrictions that would impede walking.
3. Receives usual care follow-up post ACS-related hospitalization.
4. Reported access to any computer device that has a USB port and this computer is connected to the Internet to allow upload of data from the accelerometer, and has speaker or headphones to enable listening to the intervention on the computer device of choice.
5. Reported ability to read and speak French.

Exclusion Criteria:

1. Reported sufficient physical activity during 6 months prior to hospitalization: performed at least 150 minutes of moderate-intensity physical activity per week (30 minutes five days a week) or at least 75 minutes per week of vigorous-intensity physical activity (25 minutes three days a week).
2. Indicated in the medical chart or reported by staff, physical or psychological/cognitive that would make it impossible for the patient to provide informed consent.
3. Documented New York Heart Association Class III to IV heart failure.
4. Involved in other intensive regular clinical follow-up during TAVIEenM@RCHE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2017-10-29 (Actual); Study Completion 2017-10-29 (Actual)

PRIMARY OUTCOMES:
Change in accelerometer measured steps per day | Baseline, and 12 weeks

SECONDARY OUTCOMES:
Change in accelerometer measured steps per day | Baseline, and 5 weeks
Change in self-reported energy expenditure in walking | Baseline, 5 weeks, and 12 weeks
Change in self-reported energy expenditure in moderate to vigorous physical activity | Baseline, 5 weeks, and 12 weeks

OTHER OUTCOMES:
Self-reported perceived autonomy support | 5 weeks
Change in self-reported controlled motivation | Baseline, and 5 weeks
Change in self-reported autonomous motivation | Baseline, and 5 weeks
Change in self-reported perceived competence | Baseline, and 5 weeks
Change in self-reported barrier self-efficacy | Baseline, and 5 weeks
Self-reported global quality of life | 12 weeks
Self-reported emotional quality of life | 12 weeks
Self-reported physical quality of life | 12 weeks
Self-reported social quality of life | 12 weeks
Self-reported smoking abstinence | 12 weeks
Self-reported optimal medication use | 12 weeks
Self-reported uptake in a secondary prevention program | 12 weeks
Emergency department visits identified by medical chart review | 12 weeks
Hospitalizations identified by medical chart review | 12 weeks
Self-reported angina frequency | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Cossette, Ph.D., Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Insitute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Kayser JW, Cossette S, Alderson M. Autonomy-supportive intervention: an evolutionary concept analysis. J Adv Nurs. 2014 Jun;70(6):1254-66. doi: 10.1111/jan.12292. Epub 2013 Nov 27. PMID 24279721
- [Background] Kayser JW, Cossette S, Cote J, Bourbonnais A, Purden M, Juneau M, Tanguay JF, Simard MJ, Dupuis J, Diodati JG, Tremblay JF, Maheu-Cadotte MA, Cournoyer D. Evaluation of a Web-Based Tailored Nursing Intervention (TAVIE en m@rche) Aimed at Increasing Walking After an Acute Coronary Syndrome: A Multicenter Randomized Controlled Trial Protocol. JMIR Res Protoc. 2017 Apr 27;6(4):e64. doi: 10.2196/resprot.6430. PMID 28450272